CLINICAL TRIAL: NCT04207294
Title: Bioavailability of Vitamin D-enriched Pork and Chicken in Comparison to a Vitamin D Supplement in Healthy Adults: an Acute Study
Brief Title: Vitamin D Enriched Meat Project (Acute Study)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Ulster (Other)
Collaborators: Devenish Nutrition, Lagan House, 19 Clarendon Road, Belfast, BT1 3BG (Unknown); Agri-Food and Biosciences Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: REC/19/0040
Record Dates: First submitted 2019-12-18; First posted 2019-12-20 (Actual); Last update posted 2021-06-14 (Actual); Status verified 2021-06

CONDITIONS: Vitamin D Deficiency
Keywords: Vitamin D; Pork; Chicken; Bioavailability; 25 hydroxyvitamin D; Adults; RCT; Crossover
MeSH Terms: conditions — Vitamin D Deficiency

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Vitamin D-enriched pork (Experimental): One portion of Vitamin D-enriched pork
  Interventions: Other: Pork arm
- Control pork (Placebo Comparator): One portion of control pork
  Interventions: Other: Pork arm
- Vitamin D supplement (Active Comparator): Equivocal dose of Vitamin D supplement
  Interventions: Other: Pork arm
- Vitamin D-enriched chicken (Experimental): One portion of Vitamin D-enriched chicken
  Interventions: Other: Chicken arm
- Control chicken (Placebo Comparator): One portion of control chicken
  Interventions: Other: Chicken arm

INTERVENTIONS:
Other: Pork arm — The effect of 1 portion of vitamin D-enriched pork on 25(OH)D concentration in comparison to a vitamin D supplement and control pork.
  Arms: Control pork; Vitamin D supplement; Vitamin D-enriched pork
Other: Chicken arm — The effect of 1 portion of vitamin D-enriched chicken on 25(OH)D concentration in comparison to control chicken.
  Arms: Control chicken; Vitamin D-enriched chicken

SUMMARY:
The importance of achieving an adequate vitamin D status is widely recognised, with public health and research communities heightening their interest over recent years.

Whilst vitamin D can be synthesised following skin exposure to UV light, due to public health concerns regarding sun safety, and modern indoor lifestyles, it has become evident that endogenous synthesis may not be an effective means of maintaining an adequate vitamin D status across the year. Given the marked variation in seasonally-induced cutaneous synthesis, habitually low dietary vitamin D intakes of 2-4µg/day typically reported within nationally represented population surveys, and the generally low uptake of supplementation at the population level, it is warranted to identify alternative food-based strategies to yield greater adherence to the 10µg DRV, particularly during winter months where sunlight exposure is negligible. Commodity-based biofortification may provide an innovative and viable additional food-based approach to suboptimal vitamin D status, in combination with safe sun exposure, inclusion of natural and fortified dietary sources and/or supplementation.

Meat naturally contains vitamin D3 and 25(OH)D3, yet by manipulating feeding regimes and/ or housing environments, it is possible to improve the concentration of both metabolites in animal products. Eggs, beef and pork provide viable opportunities for the enhancement of vitamin D3 and 25(OH)D3 which contribute to an increase in total vitamin D activity (vitamin D3 + [25(OH)D3 x 5]), and therefore would be expected to positively impact vitamin D status. Albeit whilst much biofortification research has been established, less is known regarding its effectiveness at raising circulating serum 25(OH)D concentrations amongst apparently healthy adults, with the exception of some plant-based foods.

Therefore, an opportunity exists to understand the bioavailability of vitamin D-enriched pork and vitamin D-enriched chicken to increase 25(OH)D concentration.

ELIGIBILITY:
Inclusion Criteria:

* · Free-living, apparently healthy Caucasian adults

  * Aged 18-65 years at Recruitment
  * Body Mass Index (BMI) ≥18.5 and <25kg/m2
  * If consuming vitamin D supplements, willing to discontinue 4 weeks prior and for duration of study
  * Non-smokers

Exclusion Criteria:

* · Non-Caucasian adults

  * Adults <18 or >65 years at recruitment
  * Taking vitamin D supplement and not willing to discontinue vitamin D supplementation for 4 weeks prior to and for duration of study
  * Current smokers
  * Pregnant/lactating females
  * Use of tanning facilities or winter vacation planned during the intervention period to a location expected to increase cutaneous synthesis
  * Severe medical illness
  * Medications which interfere with vitamin D metabolism e.g. steroid medications (e.g. prednisone), weight loss drug orlistat (e.g. Xenical and Alli), cholesterol-lowering drug cholestyramine (e.g. Questran, LoCholest and Prevalite), seizure drugs Phenobarbital and Dilantin, anti-tuberculosis, statins or thiazide diuretics
  * Intestinal malabsorption syndrome
  * Excessive alcohol use (>14 units/ week)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2020-01-16 (Actual); Primary Completion 2020-04-10 (Actual); Study Completion 2020-04-10 (Actual)

PRIMARY OUTCOMES:
Change in vitamin D concentration | Change over 24 hours (baseline (0 hr), 1.5, 3, 6, 9, 24-hour)
  Vitamin D3, vitamin D2, 25(OH)D3, 25(OH)D2) (nmol/L) in serum/plasma

SECONDARY OUTCOMES:
Calcium serum concentrations | Monitored over 24 hours (baseline (0 hr), 1.5, 3, 6, 9, 24-hour)
  Adjusted calcium
Parathyroid hormone (PTH) concentration | Change over 24 hours (baseline (0 hr), 1.5, 3, 6, 9, 24-hour)
  Plasma levels

CONTACTS AND LOCATIONS:
Locations (1):
- Human Intervention Studies Unit, Ulster University, Coleraine, Co.Londonderry, United Kingdom

IPD SHARING:
Plan to Share IPD: No